CLINICAL TRIAL: NCT05974423
Title: Prospective Randomized Trial of Narcotic vs Non-Narcotic Pain Modulation Following a Labrum Repair
Brief Title: Randomized Trial of Narcotic vs Non-Narcotic Pain Modulation After Labrum Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Cooper Health System (Other)
Collaborators: New Jersey Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 22-193
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain, Acute; Opioid Use; Labral Tear, Glenoid
Keywords: Labrum repair; opioid consumption; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Rotator Cuff Injuries | interventions — Acetaminophen; Ibuprofen; Oxycodone

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of the following groups:
  * Group 1:
    1. Oxycodone 5 mg 1 tablet every 6 hours PRN
    2. Tylenol 1000 mg every 8 hours
    3. Ibuprofen 600 mg every 6 hours as needed for pain
  * Group 2 (Experimental Group) will not be sent home with an oxycodone prescription. They will be sent home with the following prescriptions. If this does not manage their pain, they will call the resident on call who will reach out to the PI. The PI will then electronically send in a prescription of oxycodone to their pharmacy if required. The PI or operating surgeon (co-investigators) will be available 24/7 to do this. They will be sent home with these two prescriptions:
    1. Tylenol 1000 mg every 8 hours
    2. Ibuprofen 600 mg every 6 hours as needed for pain
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control - Narcotic Prescription (Active Comparator): 1. Oxycodone 5 mg 1 tablet every 6 hours PRN
  2. Tylenol 1000 mg every 8 hours
  3. Ibuprofen 600 mg every 6 hours as needed for pain
  Interventions: Drug: Tylenol, Ibuprofen, and Oxycodone
- Experimental - Non-narcotic only (Experimental): This group will not be sent home with an oxycodone prescription. They will be sent home with the following prescriptions. If this does not manage their pain, they will call the resident on call who will reach out to the PI. The PI will then electronically send in a prescription of oxycodone to their pharmacy if required. The PI or operating surgeon (co-investigators) will be available 24/7 to do this. They will be sent home with these two prescriptions:
  1. Tylenol 1000 mg every 8 hours
  2. Ibuprofen 600 mg every 6 hours as needed for pain
  Interventions: Drug: Tylenol and Ibuprofen only

INTERVENTIONS:
Drug: Tylenol, Ibuprofen, and Oxycodone — A script for these three medications will be provided
  Other Names: Both Narcotic and Non-narcotic
  Arms: Control - Narcotic Prescription
Drug: Tylenol and Ibuprofen only — A script for only these two medications will be provided initially following surgery. Should the patient need stronger medication for adequate pain control, the on-call physician will provide a script for oxycodone
  Other Names: Non-narcotic only
  Arms: Experimental - Non-narcotic only

SUMMARY:
The purpose of this study is to determine if patients age 15 to 30 years old being treated for shoulder labrum repair and SLAP lesions have significant differences in pain levels postoperatively when treated with a combination therapy of ibuprofen, and acetaminophen compared to oxycodone. Participants will be randomly placed into either the control arm and receive scripts for non-narcotic medications (Tylenol and Ibuprofen) and opioids, or the experimental arm of the study. receiving only a prescription for the non-narcotic medications. Every patient will receive a preoperative Exparel nerve block as is the standard of care for this procedure. Both groups will fill out a pain journal for 14 days following surgery and complete a pill count at the first postoperative visit to validate the amount of pain medication documented in the pain journal.

DETAILED DESCRIPTION:
The opioid crisis has illuminated the risks of opioid use for pain management, with renewed interest in reducing opioid consumption after common orthopedic procedures. Anti-inflammatory medication is an important component of multimodal pain management for patients undergoing orthopedic surgery. Several relevant studies have inquired about the use of opioid consumption in the management of total knee arthroplasty, total hip arthroplasty, total shoulder arthroplasty as well as arthroscopic shoulder surgeries. There is currently a gap in the literature, however, regarding the use of nerve blocks preoperatively in conjunction with nonopioid pharmacology postoperatively for pain. The goal is to determine if this can reduce pain levels in patients who have undergone surgical management for shoulder labrum or SLAP lesions. Hopefully, the data we can extract will allow future physicians to decrease the number of opioids prescribed and reduce the risks of prolonging the opioid epidemic.

The United States is currently in an opioid crisis. This is a public health issue that not only is limited to the United States but is echoed by countries around the world. All physicians must be accountable for the continuation of the crisis but also must be cognizant of ways to end the issue. In 2011, the United States Food and Drug Administration reported that 50 million Americans were prescribed opioids which is close to a 100 percent increase in the amount prescribed in 2008. Similarly, during that same period, opioid overdose became the leading cause of accidental death in young adults; associated with a higher risk of postoperative death, and increased risk of falls and fractures in the elderly. Many ways have been discussed to reduce the prescription of opioids such as standardized opioid prescription protocols, limits on prescription size, and restrictions on opioid use for preoperative and nonsurgical patients. Another theater of opioid use that can be addressed is that of post-operative pain management. The contribution of the potential results of our research could greatly reduce and mitigate the number of opioids prescribed postoperatively if there is no significant difference between the groups.

This will be a prospective randomized trial. Patients will be randomly placed into either the control or experimental arm of the study. Every patient will receive Exparel as is the standard of care for this procedure.

There will be two groups in this study:

* Group 1:

  1. Oxycodone 5 mg 1 tablet every 6 hours PRN
  2. Tylenol 1000 mg every 8 hours
  3. Ibuprofen 600 mg every 6 hours as needed for pain
* Group 2 (Experimental Group) will not be sent home with an oxycodone prescription. They will be sent home with the following prescriptions. If this does not manage their pain, they will call the resident on call who will reach out to the PI. The PI will then electronically send in a prescription for oxycodone to their pharmacy if required. The PI or operating surgeon (co-investigators) will be available 24/7 to do this. They will be sent home with these two prescriptions:

  1. Tylenol 1000 mg every 8 hours
  2. Ibuprofen 600 mg every 6 hours as needed for pain

At the time of diagnosis and discussion of surgical intervention, patients will be asked if they would like to participate in this research study. Patients will be considered screen fails should they meet any exclusion criteria. They will be informed that depending on which group they are randomly assigned to, they may have different prescriptions. Should the patient be randomly assigned to the control group, they will be given the above medications. Should the patient be randomly assigned to the experimental group, they will be given the above medication scripts.

To note, for shoulder surgeries, Cooper has been using Exparel as a nerve block agent as part of the standard of care.

Day 1 after surgery: both groups will begin completing their pain journal for 14 days. We will allow two methods to complete the pain journal: REDCap or paper format. The REDCap version will be emailed to patients daily so they can complete the questions. The paper format will be available to all subjects regardless of if they complete the REDCap surveys. This will be an extra measure to ensure all days are reported and there are no issues with the REDCap.

At 2 Weeks post-op: Patients' pain levels with be assessed in the immediate post-operative period at their first follow-up visit with their respective attending physician.

The subjects will keep track of pain levels through a pain journal which they fill out daily and will bring to the first post-operative appointment. At their first post-operative visit, patients will also bring their pill bottles for a pill count in the office to validate the amount described in the pain journal.

Both groups' subject's involvement will last 2 weeks post-operation. After this 2 week visit, patients will have completed their course of the study.

The current standard of practice at Cooper for orthopedic surgeons performing this procedure is oxycodone 5mg PRN, ibuprofen 600mg every 6 hours, and acetaminophen 1000mg every 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 15 - 25 years old
* Patients with a diagnosis of a labrum tear who will undergo surgical intervention

Exclusion Criteria:

* Patients under the age of 14 years old
* Patients age 26 years or older
* Patients with a nonoperative diagnosis of a labrum tear
* Patients who elect not to undergo surgical treatment
* Patients who are on opioid medications preoperatively

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain control | 2 weeks
  The subjects will keep track of pain levels through a pain journal which they fill out daily and will bring to the first post-operative appointment. At their first post-operative visit, patients will also bring their pill bottles for a pill count in the office to validate the amount described in the pain journal.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Fedorka, MD, Principal Investigator — Cooper Hospital Orthopedic Surgery
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

REFERENCES:
- [Background] Familiari F, Huri G, Simonetta R, McFarland EG. SLAP lesions: current controversies. EFORT Open Rev. 2019 Jan 28;4(1):25-32. doi: 10.1302/2058-5241.4.180033. eCollection 2019 Jan. PMID 30800477
- [Background] Hester WA, O'Brien MJ, Heard WMR, Savoie FH. Current Concepts in the Evaluation and Management of Type II Superior Labral Lesions of the Shoulder. Open Orthop J. 2018 Jul 31;12:331-341. doi: 10.2174/1874325001812010331. eCollection 2018. PMID 30197715
- [Background] Jain A, Aniq H, Mistry A. SLAP Injury and the Superior Labrum. Semin Musculoskelet Radiol. 2022 Oct;26(5):577-584. doi: 10.1055/s-0042-1758840. Epub 2022 Dec 19. PMID 36535593
- [Background] Matsuki K, Sugaya H. Complications after arthroscopic labral repair for shoulder instability. Curr Rev Musculoskelet Med. 2015 Mar;8(1):53-58. doi: 10.1007/s12178-014-9248-5. PMID 25532917
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] O'Neill A, Lirk P. Multimodal Analgesia. Anesthesiol Clin. 2022 Sep;40(3):455-468. doi: 10.1016/j.anclin.2022.04.002. Epub 2022 Aug 2. PMID 36049874
- [Background] Elmallah RK, Chughtai M, Khlopas A, Newman JM, Stearns KL, Roche M, Kelly MA, Harwin SF, Mont MA. Pain Control in Total Knee Arthroplasty. J Knee Surg. 2018 Jul;31(6):504-513. doi: 10.1055/s-0037-1604152. Epub 2017 Jul 18. PMID 28719941
- [Background] Dada O, Gonzalez Zacarias A, Ongaigui C, Echeverria-Villalobos M, Kushelev M, Bergese SD, Moran K. Does Rebound Pain after Peripheral Nerve Block for Orthopedic Surgery Impact Postoperative Analgesia and Opioid Consumption? A Narrative Review. Int J Environ Res Public Health. 2019 Sep 5;16(18):3257. doi: 10.3390/ijerph16183257. PMID 31491863
- [Background] Hamilton TW, Athanassoglou V, Trivella M, Strickland LH, Mellon S, Murray D, Pandit HG. Liposomal bupivacaine peripheral nerve block for the management of postoperative pain. Cochrane Database Syst Rev. 2016 Aug 25;2016(8):CD011476. doi: 10.1002/14651858.CD011476.pub2. PMID 27558150
- [Background] Kaye AD, Novitch MB, Carlson SF, Fuller MC, White SW, Haroldson AR, Kaiser JA, Elkersh MA, Brunk AJ, Jeha GM, Cornett EM. The Role of Exparel Plus Meloxicam for Postoperative Pain Management. Curr Pain Headache Rep. 2020 Jan 30;24(3):6. doi: 10.1007/s11916-020-0837-2. PMID 32002676
- [Background] Blair HA. Bupivacaine/Meloxicam Prolonged Release: A Review in Postoperative Pain. Drugs. 2021 Jul;81(10):1203-1211. doi: 10.1007/s40265-021-01551-9. Epub 2021 Jul 6. PMID 34228280